CLINICAL TRIAL: NCT05624879
Title: Accelerated Resolution Therapy for Early Maladaptive Grief: A Clinical Trial
Brief Title: Accelerated Resolution Therapy for Early Maladaptive Grief
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Cindy Tofthagen, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 22-005315; R01AG077656 (NIH)
Record Dates: First submitted 2022-11-15; First posted 2022-11-22 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Grief
Keywords: Family Caregiver
MeSH Terms: interventions — Palliative Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Accelerated Resolution Therapy Group (Experimental): Primary caregivers of an immediate family member enrolled in a hospice or palliative care program will receive 4 weekly sessions of accelerated resolution therapy (ART)
  Interventions: Behavioral: Accelerated Resolution Therapy
- Information and Support Group (Active Comparator): Primary caregivers of an immediate family member enrolled in a hospice or palliative care program will receive four-time and attention matched sessions of a standardized social work intervention consisting of information and provision of emotional support.
  Interventions: Other: Information and Support

INTERVENTIONS:
Behavioral: Accelerated Resolution Therapy — A brief psychotherapeutic intervention delivered by trained therapists in a maximum of 4 sessions. Sessions will focus on providing relief from the distress related to an anticipated loss and to shift focus from distress and loss back to the relationship.
  Other Names: ART
  Arms: Accelerated Resolution Therapy Group
Other: Information and Support — 4 sessions of a standardized social work intervention. Standard of care including education and active listening.
  Arms: Information and Support Group

SUMMARY:
The purpose study is to test the effects of accelerated resolution therapy (ART) on pre-loss grief and prolonged grief disorder among older adult family caregivers (FCGs). Additionally, to better understand predictors of response to ART, and cognitive processes that occur among grieving individuals following ART.

DETAILED DESCRIPTION:
Accelerated Resolution Therapy (ART) is an evidence-based treatment for post-traumatic distress in civilians and veterans that may be useful in alleviating maladaptive grief prior to bereavement and could prevent prolonged grief disorder following bereavement. Researchers are proposing to test the efficacy of ART, a low-risk, brief therapy with a strong theoretical rationale for treatment success in maladaptive grief and supported by the promising results of a recently completed preliminary trial. Additional aims of the study are to examine changes in cognitive appraisal and integration of loss following ART using a mixed methods approach and to evaluate personal, social, and psychological factors predictors of response.

During the proposed double blinded, randomized, controlled two arm clinical trial, older adult family caregivers will receive either ART or an educational program that is matched for time and attention. Each participant will receive four sessions of either the ART intervention or the control intervention. Data collection will occur at screening/enrollment (T1), at the end of the 4-session intervention period (T2) and at 6-months (T3) and 13-months post bereavement (T4). A subgroup of 20 participants randomly assigned to ART will participate in semi-structured interviews to enhance understanding of cognitive appraisal and integration of loss.

This trial will provide critical information on the efficacy of the ART intervention as a potential first-line treatment option for pre-loss grief and preventative option for prolonged grief disorder, and contribute new information about characteristics of individuals most likely to benefit from ART.

ELIGIBILITY:
Inclusion Criteria:

* Primary caregiver of immediate family member who has a life expectancy of less than 12 months
* Score of 30 or higher on the PG-12-R, indicating clinically significant pre-loss grief
* Denial of suicidal ideation or intent, with no evidence of psychotic behavior.

Exclusion Criteria:

* Since becoming a family caregiver (FCG), they have engaged in another trauma based psychotherapeutic regimen (EMDR, prolonged exposure therapy, trauma focused cognitive behavioral therapy) that could influence response to accelerated resolution therapy (ART).
* Self-reported or clinically assessed major psychiatric disorder (e.g., bipolar disorder, schizophrenia).
* Score of > 2 on the adapted CAGE questionnaire indicating alcohol /drug dependence.
* Cognitive impairment (SPMSQ > 4 errors).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2023-11-17 (Actual); Primary Completion 2028-03-14 (Estimated); Study Completion 2028-03-14 (Estimated)

PRIMARY OUTCOMES:
Changes in pre-loss grief | Baseline, 4 weeks
  Measured by 14-item self-reported Prolonged Grief-12-Revised (PG-12-R) designed to measure the grief experience of current family caregivers of persons living with progressive disease. Total grief level scores greater than or equal to 30 indicate high levels of pre-loss grief.
Changes in prolonged grief disorder | 6 and 13 months post-bereavement
  Measured by 13-item self-reported Prolonged Grief-13-Revised (PG-13-R) designed to assess indicators of pathological grief. Total scores range from 10-50; with score >29 = prolonged grief.
Changes in clinical measure of prolonged grief disorder | 6 and 13 months post-bereavement
  Measured by 31-item Structured Clinical Interview for Prolonged Grief Disorder (SCI-P) administered by healthcare professional. Higher scores = higher complicated grief symptoms.

OTHER OUTCOMES:
Change in depression | Baseline, 4 weeks, 6 and 13 months post-bereavement
  Measured using the self-reported 9-item Personal Health Questionnaire (PHQ-9) to assess how often subjects have been bother about specific problems in the last 2 weeks. Total scores range from 0-27; with score >9 = depression.
Caregiver burden | Baseline
  Measured using the self-reported 4-item Caregiver Role Overload questionnaire. Individual statement agreement on scale of "completely" agree to "not at all". Higher responses indicate more burden.
Change in perceived stress | Baseline, 6 and 13 months post-bereavement
  Measured using the self-reported 10-item NIH toolbox Item Bank/Fixed Form v2.0 - Perceived Stress questionnaire. Score range from 26-34; with higher score indicating worse stress.
Change in physical and mental health | Baseline, 6 and 13 months post-bereavement
  Measured using the self-reported 10-item Patient-Reported Outcomes Measurement Information System (PROMIS)-Global Health questionnaire. Total score range 0-20; with higher scores indicate better health.
Pessimism | Baseline
  Measured using the self-reported 10-item Revised Life Orientation Test (LOT-R). Total score range from 0-40, with higher scores indicating more optimistic
Change in life stressors | Baseline, 6 and 13 months post-bereavement
  Measured using the self-reported 13-item Social Readjustment Rating Scale where subjects indicate Yes or No and frequency of events that have occurred or expected to occur.
Change in trauma symptoms | Baseline, 4 weeks, 6 and 13 months post-bereavement
  Measured using the self-reported 20 item PTSD Checklist for DSM-5 (PCL-5) assess subjects response to very stressful experiences within the past week. Score range from 0-80; with cut-point for PTSD of 33.
Change in social support | Baseline, 4 weeks, 6 and 13 months post-bereavement
  Measured using the self-reported 8-item NIH toolbox Item Bank v2.0 - Emotional Support questionnaire. Score range from 8-40; with higher score indicating better emotional support.
Change in anxiety | Baseline, 4 weeks, 6 and 13 months post-bereavement
  Measured using the self-reported 7-item Generalized Anxiety Disorder Scale (GAD-7) to assess anxiety symptoms is the last week. Total score range from 0-2; with score >9 = high anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Tofthagen, PhD, Principal Investigator — Mayo Clinic
Locations (4):
- United States (4):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Suncoast Hospice, Clearwater, Florida
  - Mayo Clinic Florida, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No